CLINICAL TRIAL: NCT00017329
Title: Phase II Trial of PS341 (NSC 681239) in Patients With Advanced Renal Cell Carcinoma
Brief Title: PS-341 in Treating Patients With Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068678; MSKCC-01032; NCI-3031
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-12

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Bortezomib

INTERVENTIONS:
Drug: bortezomib

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of PS-341 in treating patients who have metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of PS-341 in patients with metastatic renal cell carcinoma.
* Determine the safety of this drug in these patients.

OUTLINE: This is an open-label study.

Patients receive PS-341 IV over 3-5 seconds twice weekly for 2 weeks. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed at 2 weeks.

PROJECTED ACCRUAL: A total of 12-37 patients will be accrued for this study within 6-19 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed renal cell carcinoma

  * Metastatic disease
* Unidimensionally measurable disease
* No brain metastases

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Karnofsky 70-100%

Life expectancy:

* More than 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* ALT/AST no greater than 2.5 times upper limit of normal (ULN)

Renal:

* Creatinine no greater than 1.5 times ULN

Other:

* No pre-existing neuropathy of grade 1 or greater
* No other malignancy within the past 5 years, except completely resected basal cell skin cancer, unless treated with potentially curative therapy or at low risk for recurrence
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 4 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior biologic therapy and recovered
* No concurrent biologic therapy

Chemotherapy:

* No prior cytotoxic therapy
* No concurrent cytotoxic therapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* At least 4 weeks since prior major surgery

Other:

* No other concurrent anticancer therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-04; Primary Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Drucker, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States